CLINICAL TRIAL: NCT04688502
Title: The Effects of Wearing a Face Mask During COVID-19 on Performance and Intensity Markers During CrossFit Exercise
Brief Title: Effects of Wearing a Face Mask During CrossFit Exercise
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: It was not feasible for us to run this study
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Phil Chilibeck, Professor, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2431
Record Dates: First submitted 2020-12-24; First posted 2020-12-30 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Dyspnea
MeSH Terms: conditions — Dyspnea | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- high intensity interval training wearing a face mask (Experimental): high intensity interval training wearing a face mask
  Interventions: Other: High intensity interval training
- high intensity interval training wearing no face mask (Active Comparator): high intensity interval training wearing no face mask
  Interventions: Other: High intensity interval training
- continuous exercise training wearing a face mask (Experimental): continuous exercise training wearing a face mask
  Interventions: Other: Continuous exercise training
- continuous exercise training wearing no face mask (Active Comparator): continuous exercise training wearing no face mask
  Interventions: Other: Continuous exercise training

INTERVENTIONS:
Other: High intensity interval training — High intensity interval training: 6 sets x 8 bench press, 10 pull-ups, and maximal number of box jumps (each set lasting 60 sec, with 4 minutes rest between sets)
  Arms: high intensity interval training wearing a face mask; high intensity interval training wearing no face mask
Other: Continuous exercise training — 5 pull-ups, 10 push-ups, and 15 body-weight squats, repeated for 30 minutes
  Arms: continuous exercise training wearing a face mask; continuous exercise training wearing no face mask

SUMMARY:
Face masks are important for prevention of transmission and contracting viruses such as COVID-19. Gymnasiums have been identified as being susceptible to virus transmission; therefore, wearing face masks during exercise is important during pandemics. This study will evaluate performance and physiological stress during high-intensity exercise while wearing a face mask during Crossfit exercise training.

DETAILED DESCRIPTION:
Face masks are important for prevention of transmission and contracting viruses such as COVID-19. Gymnasiums have been identified as being susceptible to virus transmission; therefore, wearing face masks during exercise is important during pandemics. This study will evaluate performance and physiological stress during high-intensity exercise while wearing a face mask during Crossfit exercise training. Twenty-four men and women will be randomly assigned to perform exercise during Crossfit exercise while wearing or not wearing a surgical face mask in a cross-over study. Two types of exercise sessions will be assessed: A high intensity interval session and a continuous exercise session. There will therefore be four exercise sessions evaluated in our randomized cross-over design: 1) high intensity exercise while wearing a face mask; 2) high intensity exercise with no face mask; 3) continuous exercise while wearing a face mask; 4) continuous exercise with no face mask. Outcome variables to be assessed include exercise performance during the sessions (total repetitions for pull-ups, push-ups, and squats during continuous exercise and total repetitions for box jumps during high-intensity exercise). Heart rate, rating of perceived exertion, and dyspnea will also be assessed throughout the exercise sessions.

ELIGIBILITY:
Inclusion Criteria:

* Experienced with CrossFit exercise training

Exclusion Criteria:

* Contra-indications to exercise as identified by a screening questionnaire (the "Get Active Questionnaire")

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-11 (Estimated); Primary Completion 2023-01-28 (Estimated); Study Completion 2023-02-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in box jumps | Up to 30 minutes
  Number of box jump repetitions during high intensity exercise
Change from baseline in pull-up, push-up, and squat repetitions | Up to 30 minutes
  Number of repetitions performed for pull-ups, push-ups, and squats

SECONDARY OUTCOMES:
Change from baseline in rating of perceived exertion | Up to 30 minutes
  Rating of perceived exertion on a scale of 1-10 (Modified Borg Scale), a higher score indicates a greater perceived exertion
Change from baseline in heart rate | Up to 30 minutes
  Heart rate (beats per minute)
Change from baseline in dyspnea | Up to 30 minutes
  Dyspnea scale (0-10), a higher score indicates increased dyspnea

CONTACTS AND LOCATIONS:
Overall Officials: Philip Chilibeck, Ph.D., Principal Investigator — University of Saskatchewan; Scotty Butcher, Ph.D., Principal Investigator — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada